CLINICAL TRIAL: NCT07401095
Title: Early Outcomes With and Without Use of a Novel Reinforced Bioinductive Implant in Arthroscopic Brostrom Repair: A Prospective Randomized Study
Brief Title: BioBrace® in Arthroscopic Brostrom Lateral Ankle Ligament Repair
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hancock Orthopedics (Other)
Collaborators: CONMED Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABBB
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: ATFL; Lateral Ankle Instability; Anterior Talofibular Ligament; Anterior Talofibular Ligament Injury; Brostrom Procedure; Brostrom; Ankle
Keywords: BioBrace; The BioBrace Implant; BioBrace Implant; ATFL; Lateral Ankle Instability; CONMED; Ankle; Ankle Injury
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Intervention Model Description: 1:1 randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control - Repair Only Group (Sham Comparator): Procedure: Standard of care Brostrom repair.
  Interventions: Other: Brostrom repair without augmentation
- BioBrace Augment Group (Experimental): Brostrom repair with BioBrace
  Interventions: Device: Brostrom repair with augmentation

INTERVENTIONS:
Device: Brostrom repair with augmentation — Brostrom repair with BioBrace
  Arms: BioBrace Augment Group
Other: Brostrom repair without augmentation — Brostrom repair without BioBrace
  Arms: Control - Repair Only Group

SUMMARY:
The purpose of this investigation is to evaluate pre- and post-operative patient reported outcomes and functional scores after an all-arthroscopic Brostrom repair using either a suture anchor construct alone or suture anchors with the BioBrace Implant.

DETAILED DESCRIPTION:
This is a single-center, prospective, randomized (1:1) interventional study investigating the use of the BioBrace® Implant in lateral ankle ligament repair procedures performed using an all-arthroscopic Broström technique. Eligible participants who meet study criteria will be enrolled and randomized into one of two study arms:

Control Group: Arthroscopic Broström repair using a suture-anchor construct only.

Treatment Group: Arthroscopic Broström repair using a suture-anchor construct augmented with the BioBrace® Implant.

Clinical evaluations will be conducted at baseline (preoperatively), and postoperatively at 1, 3, and 6 weeks, as well as at 3, 6, and 12 months using various patient-reported outcome measures to asses pain, function, activity and safety post surgery.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age at the time of surgery.
2. Able to read, understand and sign the informed consent form.
3. Willing to be available to attend each protocol required visit and complete the study required questionnaires.
4. Scheduled to undergo primary, arthroscopic Brostrom repair.

Exclusion Criteria:

1. Previous Brostrom surgery.
2. Concomitant procedures that would change the post operative course/recovery (i.e. total ankle replacement, OCD repair, foot/ankle osteotomies) as determined by the Investigator.
3. Currently participating or plans to enroll in another clinical trial during this study that would affect the outcomes of this study as determined by the Investigator.
4. History of non-compliance with medical treatment or clinical trial participation.
5. The subject is physically or mentally compromised (e.g., currently being treated for a psychiatric disorder, senile dementia, Alzheimer's disease, etc.), to the extent that the Investigator judges the subject to be unable or unlikely to remain compliant with protocol required follow-up.
6. Females of child-bearing potential who are either pregnant or breastfeeding or plan to become pregnant during the course of the study.
7. Any comorbidity or condition that renders the patient a poor surgical candidate as determined by the Investigator.
8. Hypersensitivity to any investigational device materials including collagen of animal origin (bovine type-I), poly-L-lactic acid (PLLA) or polyethylene glycol (PEG)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-08 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
American Orthopedic Foot and Ankle Society score (AOFAS) | Baseline, 1, 3, and 6 weeks & 3, 6, and 12 months
  The AOFAS Score is a clinician-based assessment tool that evaluates pain, function, and alignment in patients with foot and ankle disorders. It provides a composite score ranging from 0 to 100, with higher scores indicating better function. The system includes region-specific scales (e.g., ankle-hindfoot, midfoot, hallux) and combines both patient-reported symptoms and objective clinician findings
Foot Function Index (FFI) | Baseline, 1, 3, and 6 weeks & 3, 6, and 12 months
  The Foot Function Index (FFI) is a patient-reported questionnaire used to assess how foot conditions affect pain, disability, and activity limitation. It includes 23 items rated on a 0-10 scale, with higher scores indicating greater impairment in foot function.
Visual Analog Scale (VAS) | Baseline, 1, 3, and 6 weeks & 3, 6, and 12 months
  The Visual Analog Scale (VAS) is a tool used to measure the intensity of pain or other subjective symptoms. It consists of a 10-cm line labeled "no pain" at one end and "worst imaginable pain" at the other; patients mark their pain level on the line, which is then measured to provide a numerical score from 0 to 100.
Karlsson-Peterson score | Baseline, 1, 3, and 6 weeks & 3, 6, and 12 months
  The Karlsson-Peterson Score is a functional ankle assessment tool that evaluates symptoms such as pain, swelling, instability, stiffness, stair-climbing ability, running ability, work/activity level, and need for support, producing a total score up to 100, with higher scores indicating better ankle function.

CONTACTS AND LOCATIONS:
Locations (1):
- Hancock Orthopedics, Greenfield, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided